CLINICAL TRIAL: NCT04793893
Title: Treatment of Residual Hypermetropic Refraction on Young Patients After LASIK Using Human Fresh Corneal Lenticule Implantation Using Relex Smile Surgery
Brief Title: Treatment of Residual Hypermetropic Refraction on Young Patients After LASIK Using Human Fresh Corneal Lenticule Implantation With ReLEX Smile Surgery
Acronym: Relex-Smile
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Eye Hospital Pristina Kosovo (Other)
Responsible Party: Principal Investigator, Dr. Faruk Semiz, Head of Ophthalmology Department, Eye Hospital Pristina Kosovo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPristinaHospital
Record Dates: First submitted 2021-03-05; First posted 2021-03-11 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Refractive Errors
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment of residual hypermetropia refraction after LASIK (Experimental): The main problem at young patients post - LASIK after one year is residual hypermetropic refractive errors (especially accommodation problem) The method used in Eye Hospital is treatment with implantation of human fresh corneal lenticule (min. -1.50D) taken from myopic patients in post - LASIK patients with residual hypermetropic refractive error (min. +1.0D).
  The flap of LASIk is lifted,cleaned and then the lenticule gently inserted.The lenticule was positioned according the K2 values when is astigmatism residual refractive error.In cases where is not astigmatism the lenticule was positioned in central position under the flap.
  Interventions: Device: ReLex Smile

INTERVENTIONS:
Device: ReLex Smile — With the ReLex Smile the optical zone (lenticule diameter) and cap diameter are 6.5 and 7.5 mm respectively. After dissection of both anterior and posterior planes, the lenticule is extracted through 120 degree superior 3.5 mm incision and marked with a sterile marker (ViscotMedster).

SUMMARY:
LASIK (laser-assisted in situ keratomileusis) is a type of refractive surgery for correction of myopia, hyperopia and astigmatism. Yet approximately 30% of operated patients have symptoms like glare, halos, dry eyes and especially residual hypermetrop refractive errors.

Residual hypermetrop refractive errors are difficult to treat surgically, the current treatment is Refractive Lens Implantation - risks are similar to those of cataract surgery (endophthalmitis, loss of accommodation, etc.)

DETAILED DESCRIPTION:
The main problem at young patients post - LASIK after one year is residual refractive errors.

The method used in Eye Hospital is treatment with implantation of human fresh corneal lenticule (min. -1.50D) taken from myopic patients in post - LASIK patients with residual refractive error (min. +1.0D).

1. The flap of LASIK is lifted, cleaned and then the lenticule is gently inserted. The fresh myopic lenticule is implanted under the guidance of corneal topography in young patients with hypermetropic astigmatism residual refraction, according to the low K value. In cases where astigmatism is not present the lenticule is positioned in central position under the flap.
2. The flap of LASIK is not touched or lifted but using VisuMax femtosecond laser we created the stromal pocket with diameter 8.0 mm (1 mm larger than the optical zone of the donor lenticule) and cap thickness set to 140 μm from corneal surface and 4 mm superior incision. Hinge position flap was set at 90° angle 50° and width 4 mm, side cut angle 90°. The pocket was dissected using a blunt spatula washed with normal saline. The lenticule was held with lenticule forceps and gently inserted into the pocket through the 4 mm superior incision.

ELIGIBILITY:
Inclusion Criteria:

* residual hypermetropic refraction,
* low visual acuity

Exclusion Criteria:

* active anterior segment pathology,
* glaucoma,
* retinae detachment,

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01-08 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2025-11-08 (Estimated)

PRIMARY OUTCOMES:
Increase of visual acuity | 12 months
  Increase of visual acuity by reducing residual hypermetropy refractive errors using ReLex Smile (human fresh lenticule implantation) after LASIK.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital Pristina, Pristina, Kosovo

IPD SHARING:
Plan to Share IPD: No